CLINICAL TRIAL: NCT03639545
Title: The Effects of Empagliflozin on Functional and Structural Arterial Wall Characteristics
Brief Title: The Effects of Empagliflozin on Arterial Wall Characteristics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Mojca Lunder, MD, PhD, Research assistant at the Department of Endocrinology, Diabetes and Metabolic Diseases, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGE-SGLT2
Record Dates: First submitted 2018-08-10; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Vascular Stiffness; Hypoglycemic Agents; Diabetes Complications; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus, Type 1 | interventions — empagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- *empagliflozin* (Active Comparator): empagliflozin 25 mg daily for 12 weeks, once daily, by mouth
  Interventions: Drug: Empagliflozin 25mg
- *metformin* (Active Comparator): metformin 2000 mg daily for 12 weeks, once daily, by mouth
  Interventions: Drug: Metformin
- *empagliflozin/metformin* (Active Comparator): empagliflozin 25 mg daily and metformin 2000 mg daily for 12 weeks, by mouth
  Interventions: Drug: Empagliflozin 25mg; Drug: Metformin; Drug: Empagliflozin/Metformin
- *placebo* (Placebo Comparator): placebo for 12 weeks, once daily with water, by mouth
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Empagliflozin 25mg — The patients receive empagliflozin (25 mg daily) for 12 weeks.
  Other Names: empagliflozin
  Arms: *empagliflozin*; *empagliflozin/metformin*
Drug: Metformin — The patients receive metformin (2000 mg daily) for 12 weeks.
  Arms: *empagliflozin/metformin*; *metformin*
Drug: Empagliflozin/Metformin — The patients receive empagliflozin 25 mg daily and metformin 2000 mg daily or placebo for 12 weeks.
  Other Names: empagliflozin and metformin
  Arms: *empagliflozin/metformin*
Drug: Placebos — The patients receive for 12 weeks.
  Other Names: placebo
  Arms: *placebo*

SUMMARY:
Introduction: Diabetes mellitus is characterized by impaired arterial function and high incidence of cardiovascular events. Metformin and most recent antidiabetic groups of drugs, SGLT2 inhibitors, were in previous studies shown to reduce cardiovascular events. Until now, direct effect of empagliflozin on arterial function and its comparison to metformin was not studied yet.

Aim: The aim of the present study is to explore and compare potential direct effects of empagliflozin and metformin on arterial functional and structural arterial wall characteristics in patients with type 1 diabetes mellitus.

Methods: Patients with type 1 diabetes mellitus are randomized into four groups: 1) empagliflozin (25 mg daily), 2) metformin (2000 mg daily), 3) combination (empagliflozin 25 mg daily and metformin 2000 mg daily) and 4) control (placebo). At inclusion and after 12 weeks treatment, arterial function is assessed: endothelial function (brachial artery flow-mediated dilation (FMD), reactive hyperemia index (RHI)) and arterial stiffness (carotid pulse wave velocity (PWV), carotid-femoral PWV (cfPWV) and common carotid artery stiffness (β-stiffness)).

DETAILED DESCRIPTION:
Introduction: Diabetes mellitus is characterized by impaired arterial function and high incidence of cardiovascular events. Metformin and most recent antidiabetic groups of drugs, SGLT2 inhibitors, were in previous studies shown to reduce cardiovascular events. Until now, direct effect of empagliflozin on arterial function and its comparison to metformin was not studied yet.

Aim: The aim of the present study is to explore and compare potential direct effects of empagliflozin and metformin on arterial functional and structural arterial wall characteristics in patients with type 1 diabetes mellitus.

Methods: Patients with type 1 diabetes mellitus are randomized into four groups: 1) empagliflozin (25 mg daily), 2) metformin (2000 mg daily), 3) combination (empagliflozin 25 mg daily and metformin 2000 mg daily) and 4) control (placebo). At inclusion and after 12 weeks treatment, arterial function is assessed: endothelial function (brachial artery flow-mediated dilation (FMD), reactive hyperemia index (RHI)) and arterial stiffness (carotid pulse wave velocity (PWV), carotid-femoral PWV (cfPWV) and common carotid artery stiffness (β-stiffness)).

Background:

Diabetes mellitus is characterized by chronic hyperglycaemia causing chronic microvascular and macrovascular complications. Among the microvascular complications, diabetic retinopathy, neuropathy and nephropathy are included. Macrovascular complications include atherosclerotic brain-vascular disease, coronary disease and peripheral arterial disease. Chronic complications of diabetes pose a greater risk of disability, development of blindness, renal failure, neuropathy and cardiovascular disease. Consequently, a good glycemic control is crucial to protect the patients from the development of chronic complications. In this regard, glycemic control is of primary importance, as well as the choice of treatment that can further improve the functioning of the arteries and thus protect against the onset of cardiovascular damage or complications.

For the treatment of hyperglycemia patients with type 1 diabetes need insulin. Some oral anti-diabetics have been found to improve glycemic control, reduce insulin consumption (the total daily insulin dose), and also protect against the development of cardiovascular complications. Such effects have been shown in clinical studies for metformin. The latter improved from endothelium-dependent relaxation of the arteries and reduced insulin resistance, but most studies were performed in patients with type 2 diabetes and studies in type 1 diabetes are limited.

A novel group of oral antidiabetics are SGLT2 inhibitors, such as empagliflozin, reduce glucose reabsorption in proximal kidney tubules and increase glucose excretion through urine. Most of the previous studies on the efficacy of empagliflozin basic antidiabetic activity and additional effects have been performed in patients with type 2 diabetes. They were shown to improve glyceamia control and also reduced blood pressure body weight. In patients with type 1 diabetes, favorable effects of empagliflozin on the reduction of arterial wall stiffness and blood pressure reduction were observed, but no systematic studies were performed yet and the mechanisms behind the beneficial effects are not known yet.

Methods:

Type 1 diabetes mellitus patients are being recruited. The patients are equally randomized into 4 groups that receive one of the three drugs in addition to insulin. The groups were as follows: 1) empagliflozin group (receiving 25 mg daily), 2) metformin group (receiving 2000 mg daily), combination group (receiving empagliflozin 25 mg daily and metformin 2000 mg daily) and 4) control group (receiving placebo). The duration of the study period is 12 weeks. All subjects are voluntarily participating in this study. The study was approved by the National Medical Ethics Committee of Slovenia.

At the beginning of the study, a complete history and full medical examination of each patient are performed. At inclusion to the study and after 12 weeks of treatment, arterial function measurements are performed, comprising of i) measurements of endothelial function (brachial artery flow-mediated dilation (FMD), reactive hyperemia index (RHI)); and ii) measurements of arterial stiffness (carotid artery pulse wave velocity (PWV), carotid-femoral PWV (cfPWV) and common carotid artery stiffness (β-stiffness)). Additionally, venous blood samples are obtained at the beginning and at the end of the study period. Automated sphygmomanometer is used for blood pressure measurements. Ultrasound measurements are obtained on Aloka ProSound alpha7 machine with integrated high resolution eTracking system. Endothelial function, by means of brachial artery FMD, was assessed in accordance to the current guidelines. Reactive hyperemia index is measured using Endopat 2000 device (Itamar Medical Ltd., Caesarea, Israel), while cfPWV is obtained using SphygmoCor device (AtCor Medical, Sydney, Australia) with SphygmoCor CvMS software (version 9).

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 1

Exclusion Criteria:

* diagnosed advanced heart, kidney or liver failure
* benign prostatic hyperplasia
* prostatic carcinoma
* frequent urinary tract infections
* non-type 1 diabetes mellitus

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Arterial function | the change of arterial function from baseline to 12 weeks of treatment
  Endothelial function and arterial stiffness will be measured.

SECONDARY OUTCOMES:
Glycemic control | the change of HbA1c from baseline to 12 weeks of treatment
  HbA1c will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, prof, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lunder M, Janic M, Japelj M, Juretic A, Janez A, Sabovic M. Empagliflozin on top of metformin treatment improves arterial function in patients with type 1 diabetes mellitus. Cardiovasc Diabetol. 2018 Dec 3;17(1):153. doi: 10.1186/s12933-018-0797-6. PMID 30509271